CLINICAL TRIAL: NCT04676906
Title: A Phase 0, Open-label, Candidate Selection Study Assessing the Pharmacokinetics of 3 Drug Candidates After a Single Intravenous, 14C-labelled Microdose in Healthy Male Subjects
Brief Title: A Study Investigating the Distribution and Metabolism of Three 14C-labeled Radioactive Study Compounds
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NN9520-4709; 2020-003449-13 (Registry Identifier: European Medicines Agency (EudraCT)); U1111-1255-1447 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-12-01; First posted 2020-12-21 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study compound 1 (Experimental): Up to 6 volunteers will receive one dose of study compound 1
  Interventions: Drug: NNC0113-6861
- Study compound 2 (Experimental): Up to 6 volunteers will receive one dose of study compound 2
  Interventions: Drug: NNC0113-6860
- Study compound 3 (Experimental): Up to 6 volunteers will receive one dose of study compound 3
  Interventions: Drug: NNC0113-6891

INTERVENTIONS:
Drug: NNC0113-6861 — Study compound 1 - Each participant will receive a single intravenous (i.v) dose of [14C]-NNC0113-6861
  Arms: Study compound 1
Drug: NNC0113-6860 — Study compound 2 - Each participant will receive a single i.v dose of [14C]-NNC0113-6860
  Arms: Study compound 2
Drug: NNC0113-6891 — Study compound 3 - Each participant will receive a single i.v dose of [14C]-NNC0113-6891
  Arms: Study compound 3

SUMMARY:
People with type 2 diabetes have too much sugar in their blood and need treatment to control their sugar level. The 3 study compounds in this study are similar to an approved antidiabetic medicine that helps to lower blood sugar levels in people with type 2 diabetes. This approved antidiabetic medicine is generally safe and well tolerated. The study compounds are expected to have the same antidiabetic effect as the approved medicine. The purpose of this study is to investigate how quickly and to what extent each of the 3 study compounds are broken down in the body (this is called pharmacokinetics). The dose of each study compound will be very low (this is called a microdose), and will be labelled with a small amount of carbon-14. This is radioactive, and it makes it possible to track the study compound in the blood. The 3 study compounds in this study have not been given to humans before. The study will be performed in up to 18 healthy male volunteers. The study will consist of 3 groups of 6 volunteers each. Each participant will receive only one dose of study medicine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject.
* Sex : Male.
* Age 18 to 54 years, inclusive, at the time of signing informed consent.
* Body mass index (BMI) 18.0 to 30.0 kg/m^2, inclusive, at the time of signing informed consent .

Exclusion Criteria:

* Known or suspected hypersensitivity to study product(s) or related products.
* Any disorder that in the Investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol.
* Glycosylated haemoglobin (HbA1c) equal to or above 6.5% (48 mmol/mol) at screening.
* Personal or first-degree relative(s) history of multiple endocrine neoplasia Type 2 or medullary thyroid carcinoma.
* Subjects with a history of malignant neoplasms within the past 5 years prior to screening.
* Presence or history of pancreatitis (acute or chronic; as declared by the subject or reported in the medical records).
* Participation in a study with a radiation burden of above 0.1 millisievert (mSv) in the period of 1 year prior to screening.

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
The apparent elimination half-life of each of the 3 study compounds and their active metabolite after a single iv dose of each of the 3 study compounds | From time of first dosing (Day 1) until Day 64
  hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency ( dept. 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com